CLINICAL TRIAL: NCT05435209
Title: A Longitudinal Cohort Study to Assess Effectiveness and B-memory Response to the Quadrivalent HPV Vaccine 9 Years Post-vaccination Among HIV-Infected Boys and Girls Ages 9-14 Years in Kenya
Brief Title: Effectiveness of the Q-HPV Vaccine 9-years Post Vaccination Among HIV Positive Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Nelly Mugo, Associate Professor, School of Medicine: Global Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00013326
Record Dates: First submitted 2022-06-10; First posted 2022-06-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: HPV Infection; HPV Vaccination
Keywords: Genital HPV infection; quadrivalent HPV vaccination; HIV-infected; adolescents
MeSH Terms: conditions — Papillomavirus Infections | interventions — Vaccines, Synthetic

STUDY DESIGN:
Intervention Model Description: Quadrivalent HPV vaccine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Quadrivalent HPV Vaccine (Experimental): Gardasil® 0.5 mL administered intramuscularly in the deltoid or anterolateral area of the thigh
  Interventions: Drug: Quadrivalent Human Papillomavirus (Types 6,11,16,18) Recombinant Vaccine

INTERVENTIONS:
Drug: Quadrivalent Human Papillomavirus (Types 6,11,16,18) Recombinant Vaccine — Gardasil
  Other Names: Gardasil-4

SUMMARY:
The risk for Human Papillomavirus (HPV) infection persists through an individual sexual life and duration of protection is critical to vaccine effectiveness in protection from oncogenic hrHPV infection. HIV-infected individuals have an increased risk for HPV infection, and persistent infection.

Most vaccine efficacy data among HIV-infected adolescents is represented by immunogenicity data, and there is little published literature on vaccine effectiveness as assessed by persistent incident genital HPV infection.

Investigators shall re-enroll a cohort of previously vaccinated HIV-infected girls and boys for assessment of genital HPV infection 9-years post initial 3 doses of vaccination with quadrivalent HPV vaccine at ages 9 to 14 years.

DETAILED DESCRIPTION:
Background: Genital Human Papilloma Virus (HPV) infections occur rapidly after sexual debut, and immunosuppressed individuals are at greater risk for incident and persistent infection. HPV vaccine contains virus-like particles (VLP), which are highly immunogenic and induce a robust humoral response that has been demonstrated to confer long term protection from HPV infection and associated disease among HIV-uninfected individuals. The magnitude of type-specific vaccine induced neutralizing HPV antibody responses are diminished among HIV-infected compared to uninfected individuals.

There is no established minimum level of antibody that predicts protection against HPV infection or associated disease, the impact of lower antibody titers among HIV infected individuals on vaccine efficacy is unknown. The risk of HPV exposure persists throughout a person's sexual life and the duration of protection, especially when the vaccine is given in the early adolescent period is critical to vaccine effectiveness. Long lasting memory is characterized by memory B cells and long-lived plasma cells and a QHPV booster dose has demonstrated an anamnestic response among HIV-infected adolescents.

HPV efficacy and effectiveness data for HIV-uninfected individuals has informed the current World Health Organization (WHO) two-dose vaccine schedule. The field lacks data on effectiveness of three dose or two-dose for the HIV-infected adolescents. The current on-going research for single dose schedules gives urgency to the determination of long-term efficacy of three HPV vaccine 231 doses for the HIV-infected adolescent.

Investigators shall recall HIV-infected girls and boys who were previously vaccinated at ages 9-14 years with three doses of the quadrivalent vaccine (QHPV) in 2014 and evaluated for vaccine immunogenicity.

Method: The participants will be assessed for genital warts and genital HPV infection. Type specific HPV DNA will be assessed using genital swabs and genital warts assessed through physical examination among sexually active participants at enrollment, month 6 &12.

Among those that have not become sexually active, or that decline a genital exam, a self-collected swab will be requested. A sub-set of approximately 30 participants, will receive a booster dose of QHPV, from this subset, Peripheral Blood Mononuclear Cells (PBMC) and plasma samples will be collected at enrollment, at month 1 and month 12 to evaluate for memory B and T cell responses.

The total duration of study follow up will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* enrolled previously and received received three doses of quadrivalent HPV- vaccine in 2014

Exclusion Criteria:

* Decline re-enrollment
* unable to provide informed consent
* minor without parent or guardian consent

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 158 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Persistent Genital HPV infection | Nine years after primary vaccination
  Number of participants with incident persistent genital infection with the QHPV specific serotypes: -6, -11, -16 and -18 and additional 13 oncogenic HPV serotypes (31,33,35,39,45,51,52,56,58,59,66, 68,73)
Sustained QHPV vaccine specific antibody titers | Nine years after primary vaccination
  Concentration of QHPV specific antibody titers (HPV -6, -11, -16 & -18) nine years after primary vaccination

SECONDARY OUTCOMES:
Immune memory following three doses of QHPV | One month after booster vaccine
  B cell marker concentration following a booster 4th dose of QHPV

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mugo, MD, Principal Investigator — University of Washington
Locations (1):
- Phrd-Ccr-Kemri, Thika, Kiambu County, Kenya